CLINICAL TRIAL: NCT05726682
Title: A Phase 2, Single Arm, Multicohort, Open Label, Multicenter Trial of Off-the-shelf Natural Killer (NK) Cells (SAR445419) in Patients With High-risk Myeloid Malignancies Undergoing Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: A Study to Investigate Use of Off-the-shelf Natural Killer (NK) Cells (SAR445419) in Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to cancel trial, not related to safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT17550; U1111-1275-1345 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-02-02; First posted 2023-02-14 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Allogenic Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: This is a parallel multicohort, phase 2, single-arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- High risk AML and MDS (Experimental): Participants with high risk acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) undergoing allogeneic HSCT will receive 3 doses of SAR445419. A myeloablative conditioning (MAC) and a reduced intensity conditioning (RIC) cohort will be included.
  Interventions: Drug: SAR445419

INTERVENTIONS:
Drug: SAR445419 — Pharmaceutical form: cell suspension Route of administration: Intravenous (IV) injection

SUMMARY:
This is a multicenter, parallel multicohort, phase 2, single-arm study for adjunctive treatment in participants with high-risk myeloid malignancies undergoing allogeneic HSCT. The purpose of this study is to assess the safety and preliminary efficacy of off-the-shelf (OTS) ex vivo expanded NK cells (SAR445419) in improving relapse free survival (RFS).

DETAILED DESCRIPTION:
The expected duration of the study for a participant is about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 (Cohort A - MAC) or 18-75 (Cohort B - RIC)
* Participants with high-risk AML/MDS who are scheduled to undergo stem cell transplantation with matched sibling donor (MSD), matched unrelated donor (MUD) or haploidentical donor sourced HSCT
* Hematopoietic Cell Transplantation Comorbidity Index (HCT-CI) ≤ 3 (cohort A / MAC participants only)
* Adequate major non-hematopoietic organ system function
* Karnofsky performance score ≥70%
* Body weight ≥45 kg

Exclusion Criteria:

* AML beyond CR1
* Presence of FLT3 mutations
* Uncontrolled bacterial, viral, or fungal infections at time of enrollment
* Positive test for human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS)
* Positive hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating acute or chronic infection
* Diagnosis of prior immunodeficiency or organ transplantation requiring immunosuppressive therapy
* Active or chronic autoimmune condition requiring systemic immunosuppressive or immunomodulatory therapy
* Prior allogeneic transplantation
* HSCT graft DSA ≥3000 MFI
* Current use of systemic corticosteroids at physiologic doses ≤ 0.2 mg/kg/day of prednisone or equivalent
* Use of checkpoint inhibitor therapy within 4 weeks prior to the start of HSCT conditioning regimen The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2027-02-12 (Estimated); Study Completion 2027-10-11 (Estimated)

PRIMARY OUTCOMES:
Rate of relapse free survival (RFS) post allogeneic hematopoietic stem cell transplantation (HSCT) | 12 months post HSCT
  Percentage of patients who are relapse free and alive at 12 months from the date of HSCT and who received at least the first 2 planned doses of SAR445419
Frequency of cytomegalovirus (CMV) reactivation/infection in CMV seronegative participants who receive a CMV seronegative HSCT graft | From baseline up to 2 years
Frequency of life-threatening (grade 4) infusion related reactions (IRR) or cytokine release syndrome (CRS) that does not resolve to grade 1 within 72 hours despite therapy | From baseline up to 2 years
Frequency of life threatening (grade 4) tumor lysis syndrome (TLS) | From baseline up to 2 years
Frequency of life-threatening (grade 4) immune cell-associated neurotoxicity syndrome (ICANS) that does not resolve to grade 1 within 72 hours despite therapy | From baseline up to 2 years
Frequency of grade 3-4 acute graft versus host disease (aGVHD) | From baseline up to 2 years
Frequency of non-relapse mortality (NRM) | 100 days post HSCT
Frequency of graft failure | 100 days post HSCT
  Frequency of primary or secondary graft failure
Frequency of overall mortality | 100 days post HSCT

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) | From baseline up to 2 years
  AEs characterized by type and severity as graded by the national cancer institute common terminology criteria for adverse events (NCI CTCAE) v.5.0, timing, seriousness, and relationship to study treatments. All AEs will be captured from signing of informed consent until 30 days after the last SAR445419 administration. All serious AEs (SAEs) and AEs of special interest (AESIs) will be captured until the end of the study.
Number of participants with acute Graft-Versus-Host-Disease (aGVHD) | 6, 12, 18 and 24 months post-HSCT
  The cumulative incidence of grade 2-4 and 3-4 aGVHD
Number of participants with chronic Graft-Versus-Host-Disease (cGVHD) | 6, 12, 18 and 24 months post-HSCT
  The cumulative incidence of cGVHD graded as mild, moderate or severe
Proportion of participants who are alive and do not need ongoing immune suppression to control GVHD | 6, 12, 18 and 24 months post-HSCT
Cumulative incidence of relapse | 6, 12, 18 and 24 months post-HSCT
Rate of relapse free survival (RFS) | 6, 12, 18 and 24 months post-HSCT
Rate of overall survival (OS) | 6, 12, 18 and 24 months post-HSCT
Rate of non-relapse mortality (NRM) | 6, 12, 18 and 24 months post-HSCT
Rate of GVHD-free relapse-free survival (GRFS) | 6, 12, 18 and 24 months post-HSCT
Time to hematologic recovery (platelet and neutrophil count recovery) post-HSCT | From baseline up to approximately 180 days
Frequency of donor cell engraftment | 28 and 100 days, and 6 and 12 months post-HSCT
  The proportion of patients with full chimerism (≥95% donor cells), mixed chimerism (5-95% donor cells) and graft rejection (<5% donor cells)
Frequency of primary graft failure | 28 days post-HSCT
Frequency of secondary graft failure | 100 days and 12, 18 and 24 months post-HSCT
Cumulative incidence of CMV reactivation or infection and symptomatic BK-virus (BKV) hemorrhagic cystitis | 100 days and 6 and 12 months post-HSCT
Cumulative incidence of grade 2-4 and grade 3-4 infections during the on-treatment period | Until 30 days after the last administration of SAR445419
Change from baseline in Quality of life in Acute Myeloid Leukemia (AML-QoL) score | 28 and 100 days and 6, 9 and 12 months post HSCT
  AML-QoL is a 27 item questionnaire to measure quality of life in patients with Acute Myeloid Leukemia and high-risk Myelodysplastic Syndrome, covering seven different domains and with lower scores indicating better quality of life. AML-QoL uses 5-point Likert type scale ranging from 1: "Never" to 5: "Almost always" for the 26 items included in domains and ranging from 1: "Excellent" to 5: "Poor" for the QOL item.
Change from baseline in Functional Assessment of Cancer Therapy - Bone Marrow Transplantation (FACT-BMT) score | 28 and 100 days and 6, 9 and 12 months post HSCT
  FACT-BMT is a 50 item questionnaire to measure quality of life in bone marrow transplant patients covering five different domains and with higher scores indicating better quality of life. FACT-BMT questionnaire uses likert type scale with responses measuring from 0-4 (where 0 = not at all; 1 = a little bit; 2 = somewhat, 3 = quite; and 4 = very much)
Change from baseline in Patient Global Impression of Severity (PGIS) score | 28 and 100 days and 6, 9 and 12 months post HSCT
  PGIS scale is a single-item with a self-reported categorical scale to assess patient's impression of disease severity. PGIS contains response options ranging from 0 (none) to 4 (severe).
Change from baseline in Patient Global Impression of Change (PGIC) score | 28 and 100 days and 6, 9 and 12 months post HSCT
  PGIC scale is a single item with a self-reported categorical scale designed to assess patient's impression of change in disease symptom severity. PGIC contains response options ranging from 0 (no-change) to 7 (considerable improvement).
Change from baseline in Functional Assessment of Chronic Illness Therapy GP5 question (FACIT-GP5) score | 7, 14 and 35 days post-HSCT
  FACIT-GP5 is single item to assess global side effect bother. FACIT-GP5 uses likert type scale with responses Scores range from 0 (not at all bothered by side effect) to 4 (very much bothered by side effects).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org